CLINICAL TRIAL: NCT01686334
Title: Wilms' Tumor (WT1) Antigen-targeted Dendritic Cell Vaccination to Prevent Relapse in Adult Patients With Acute Myeloid Leukemia: a Multicenter Randomized Phase II Trial
Brief Title: Efficacy Study of Dendritic Cell Vaccination in Patients With Acute Myeloid Leukemia in Remission
Acronym: WIDEA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zwi Berneman (Other)
Collaborators: Kom Op Tegen Kanker (Other); Stichting tegen Kanker (Other); Research Foundation Flanders (Other)
Responsible Party: Sponsor-Investigator, Zwi Berneman, Full Professor, University Hospital, Antwerp
Organization: University Hospital, Antwerp (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCRG12-001
Record Dates: First submitted 2012-07-26; First posted 2012-09-18 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: in complete remission; Adult (>18 years) at very high risk of relapse
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Pathologic Complete Response | interventions — lentiviral minigene vaccine of COVID-19 coronavirus

ARMS (2):
- DC vaccine (Experimental): Vaccination with autologous WT1 mRNA-electroporated DCs plus follow-up care. Patients receiving low-intensity chemotherapy are allowed to continue this treatment in combination with DC vaccination.
  Interventions: Biological: DC vaccine
- Control arm (No Intervention): Follow-up care. Patients receiving low-intensity chemotherapy are allowed to continue this treatment during the follow-up care

INTERVENTIONS:
Biological: DC vaccine — Autologous WT1 mRNA-electroporated DCs
  Arms: DC vaccine

SUMMARY:
The primary aim of this innovative immunotherapeutic study is to determine whether the antileukemic effects seen in our previous phase I/II study can be confirmed in a large cohort of patients and whether dendritic cell vaccination can significantly prevent relapse and increase survival of acute myeloid leukemia (AML) patients by eradicating minimal residual disease.

DETAILED DESCRIPTION:
Together with the Transplant Committee of the Belgian Hematological Society (BHS), we will perform a multicenter randomized open-label phase II clinical study in 130 patients with acute myeloid leukemia (AML). Adult patients (> 18 years) with AML who have entered morphological CR or CRi after (1) intensive chemotherapy (i.e (i) at least one cycle of induction and one cycle of consolidation chemotherapy or (ii) one to two cycles of CPX-351 induction treatment and up to two cycles of CPX-351 consolidation treatment) or (2) low-intensity chemotherapy (i.e (iii) at least two cycles to maximum six cycles of hypomethylating agents whether or not combined with venetoclax or (iv) at least two cycles to maximum six cycles of low-dose cytarabine combined with venetoclax); and fulfilling all other eligibility criteria will be randomized to be vaccinated with dendritic cells or to receive regular follow-up care. After randomization, patients receiving low-intensity chemotherapy are allowed to continue this treatment in combination with DC vaccination or the follow-up care. The primary aim of this innovative immunotherapeutic study is to determine whether the antileukemic effects seen in our previous phase I/II study can be confirmed in a large cohort of patients and whether dendritic cell vaccination can significantly prevent relapse and increase survival of AML patients by eradicating minimal residual disease. Patients will be recruited at 8 different centers in Belgium. Recruitment will start in the second half of 2013 and will last for 10 years or until 130 efficacy-evaluable AML patients are included. In the interventional group, 65 patients will be treated during two years with autologous dendritic cells loaded by messenger RNA electroporation with the Wilms' tumor antigen (WT1). The dendritic cell therapy product will be generated and generally administered in the coordinating center, which is the Antwerp University Hospital, more specifically the Center for Cell Therapy and Regenerative Medicine (CCRG) and the Division of Hematology, both headed by Prof. Zwi Berneman. After inclusion of 130 efficacy-evaluable patients, relapse rate, relapse-free survival and overall survival analysis will be performed. Tumor marker levels and immune activation will also be monitored to compare the 2 groups at a molecular and immunological level. General and disease-specific quality of life will be evaluated using quality of life questionnaires at regular time points.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (AML) according to the 2008 criteria of the World Health Organization (WHO).

  * all French-American-British (FAB) subtypes, except:

    - M3 (acute promyelocytic leukemia)
  * all cases of de novo AML or secondary AML with ≥ 20 % blasts in peripheral blood and/or bone marrow, except:

    * AML secondary to myeloproliferative neoplasms (MPN)
    * AML secondary to exposure of leukemogenic agents (t-AML) unless treated with CPX-351 chemotherapy or hypomethylating agents combined with venetoclax.
* Completion of one of the following treatment options:

  * I) Intensive chemotherapy:

    * (1) at least one cycle of induction chemotherapy and one cycle of consolidation chemotherapy (low-dose cytarabine as consolidation therapy is allowed) OR
    * (2) one to two cycles of CPX-351 induction treatment and up to two cycles of CPX-351 consolidation treatment OR
  * II) Low-intensity chemotherapy:

    * (3) at least two cycles to maximum six cycles of hypomethylating agents whether or not combined with venetoclax OR
    * (4) at least two cycles to maximum six cycles of low-dose cytarabine combined with venetoclax;
  * resulting in:

    * morphological complete remission (CR), i.e. bone marrow blast count <5% with neutrophil count >1000 cells/µL and platelet count >100,000 cells/µL OR
    * morphological complete remission with incomplete blood recovery (CRi), i.e. bone marrow blast count <5% with neutrophil count <1000 cells/µL or platelet count <100,000 cells/µL.

For the purpose of this study protocol, platelet count must be >50,000 cells/µL.

* Adult (≥ 18 years) at very high risk of relapse according to:

  * Age ≥ 60 years, and/or
  * Adverse biological features (e.g. adverse cytogenetics, adverse morphological features, adverse molecular features, hyperleukocytosis (> 100000 cells/µL)), and
  * Ineligible for or unwilling to receive hematopoietic stem cell transplantation.
* WHO performance status: grade 0, 1 or 2 at the time of enrollment. For definition of performance status, see: http://www.ecog.org/general/perf_stat.html
* Absence of any psychological, familial, sociological, geographical or physical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before study entry.

Exclusion Criteria:

* Participation in any other interventional clinical trial during the study period.
* History or concomitant presence of any other malignancy, except for:

  * non-melanoma skin cancer
  * carcinoma in situ of the cervix
  * any other effectively treated malignancy that has been in remission for >5 years or that is highly likely to be cured at the time of enrollment.
* Concomitant presence of any immunosuppressive disease (e.g. HIV) or any active autoimmune condition, except for vitiligo.
* Concomitant use of systemic corticosteroids in immunosuppressive doses (>1 mg/kg/day of prednisone, or equivalent dose for other corticosteroid preparations) or any other immunosuppressive agent. A minimum of 4 weeks must have elapsed between the last dose of immunosuppressive therapy and the first vaccination. Topical corticosteroids are permitted, except if applied at the sites of DC injection.
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2012-10; Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | At study completion, an average of 5 year
  The primary objective of this randomized phase II clinical study is to determine the effect of WT1-targeted dendritic cell vaccination on overall survival in adult AML patients at very high risk of relapse and in complete remission.

SECONDARY OUTCOMES:
Relapse rate | At study completion, an average of 5 year
  to determine the effect of WT1-targeted dendritic cell vaccination on relapse rate in adult AML patients at very high risk of relapse and in complete remission.
relapse-free survival | At study completion, an average of 5 year
  to determine the effect of WT1-targeted dendritic cell vaccination on relapse-free survival in adult AML patients at very high risk of relapse and in complete remission.
Change in WT1 mRNA levels in peripheral blood | Through study completion, at every vaccination during 2 years
  Efficacy assessment will also be performed on a molecular level. To this end, peripheral blood samples will be obtained from participants in both study groups (vaccine group and control group) and analyzed by qRT-PCR for WT1 expression, which is a promising molecular biomarker in AML.
Immune activation | After the 4th DC vaccine
  This study aims to examine the presence of leukemia-specific immune responses in AML patients in remission and to investigate whether they can be induced or increased in these patients by WT1 mRNA-electroporated DC vaccination.
General and disease-specific quality of life | At study completion, an average of 5 year
  Patients will be asked to fill out general and disease-specific quality of life questionnaires to assess changes in general and disease-specific quality of life during the study at regular time points

OTHER OUTCOMES:
Tertiary: Safety | At study completion, an average of 5 year
  To corroborate the safety of WT1 mRNA-electroporated DC vaccination in adult patients with AML. Safety will be assessed at every visit by adverse event reporting and clinical laboratory tests.
Exploratory: Effect of low-intensity chemotherapy | At study completion, an average of 5 year
  To evaluate the effect of low-intensity chemotherapy on the primary and secondary objectives.

CONTACTS AND LOCATIONS:
Overall Officials: Zwi Berneman, MD, PhD, Study Director — University Hospital, Antwerp; Evelien LJ Smits, MSc, PhD, Principal Investigator — Universiteit Antwerpen; Sébastien Anguille, MD, PhD, Principal Investigator — University Hospital, Antwerp; Ann Van de Velde, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (8):
- Belgium (8):
  - ZNA Cadix, Antwerp
  - Antwerp University Hospital, Antwerp
  - University Hospital Brussels, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Ghent University Hospital, Ghent
  - Centre Hospitalier Universitaire de Liège, Liège
  - AZ Delta, Roeselare
  - CHU Mont Godinne, Yvoir

REFERENCES:
- [Background] Van Tendeloo VF, Van de Velde A, Van Driessche A, Cools N, Anguille S, Ladell K, Gostick E, Vermeulen K, Pieters K, Nijs G, Stein B, Smits EL, Schroyens WA, Gadisseur AP, Vrelust I, Jorens PG, Goossens H, de Vries IJ, Price DA, Oji Y, Oka Y, Sugiyama H, Berneman ZN. Induction of complete and molecular remissions in acute myeloid leukemia by Wilms' tumor 1 antigen-targeted dendritic cell vaccination. Proc Natl Acad Sci U S A. 2010 Aug 3;107(31):13824-9. doi: 10.1073/pnas.1008051107. Epub 2010 Jul 14. PMID 20631300
- [Background] Van Driessche A, Van de Velde AL, Nijs G, Braeckman T, Stein B, De Vries JM, Berneman ZN, Van Tendeloo VF. Clinical-grade manufacturing of autologous mature mRNA-electroporated dendritic cells and safety testing in acute myeloid leukemia patients in a phase I dose-escalation clinical trial. Cytotherapy. 2009;11(5):653-68. doi: 10.1080/14653240902960411. PMID 19530029
- [Background] Van Driessche A, Gao L, Stauss HJ, Ponsaerts P, Van Bockstaele DR, Berneman ZN, Van Tendeloo VF. Antigen-specific cellular immunotherapy of leukemia. Leukemia. 2005 Nov;19(11):1863-71. doi: 10.1038/sj.leu.2403930. PMID 16121214
- [Background] Van Driessche A, Berneman ZN, Van Tendeloo VF. Active specific immunotherapy targeting the Wilms' tumor protein 1 (WT1) for patients with hematological malignancies and solid tumors: lessons from early clinical trials. Oncologist. 2012;17(2):250-9. doi: 10.1634/theoncologist.2011-0240. Epub 2012 Jan 30. PMID 22291091
- [Background] Anguille S, Willemen Y, Lion E, Smits EL, Berneman ZN. Dendritic cell vaccination in acute myeloid leukemia. Cytotherapy. 2012 Jul;14(6):647-56. doi: 10.3109/14653249.2012.693744. PMID 22686130
- [Background] Anguille S, Lion E, Smits E, Berneman ZN, van Tendeloo VF. Dendritic cell vaccine therapy for acute myeloid leukemia: questions and answers. Hum Vaccin. 2011 May;7(5):579-84. doi: 10.4161/hv.7.5.14652. Epub 2011 May 1. PMID 21422813
- [Background] Smits EL, Anguille S, Cools N, Berneman ZN, Van Tendeloo VF. Dendritic cell-based cancer gene therapy. Hum Gene Ther. 2009 Oct;20(10):1106-18. doi: 10.1089/hum.2009.145. PMID 19656053
- [Background] Anguille S, Van de Velde AL, Smits EL, Van Tendeloo VF, Juliusson G, Cools N, Nijs G, Stein B, Lion E, Van Driessche A, Vandenbosch I, Verlinden A, Gadisseur AP, Schroyens WA, Muylle L, Vermeulen K, Maes MB, Deiteren K, Malfait R, Gostick E, Lammens M, Couttenye MM, Jorens P, Goossens H, Price DA, Ladell K, Oka Y, Fujiki F, Oji Y, Sugiyama H, Berneman ZN. Dendritic cell vaccination as postremission treatment to prevent or delay relapse in acute myeloid leukemia. Blood. 2017 Oct 12;130(15):1713-1721. doi: 10.1182/blood-2017-04-780155. Epub 2017 Aug 22. PMID 28830889
- [Background] Van Acker HH, Versteven M, Lichtenegger FS, Roex G, Campillo-Davo D, Lion E, Subklewe M, Van Tendeloo VF, Berneman ZN, Anguille S. Dendritic Cell-Based Immunotherapy of Acute Myeloid Leukemia. J Clin Med. 2019 Apr 27;8(5):579. doi: 10.3390/jcm8050579. PMID 31035598
- [Background] Smits EL, Stein B, Nijs G, Lion E, Van Tendeloo VF, Willemen Y, Anguille S, Berneman ZN. Generation and Cryopreservation of Clinical Grade Wilms' Tumor 1 mRNA-Loaded Dendritic Cell Vaccines for Cancer Immunotherapy. Methods Mol Biol. 2016;1393:27-35. doi: 10.1007/978-1-4939-3338-9_3. PMID 27033213
- [Background] Z. Berneman, S. Anguille, Y. Willemen, A. Van de Velde, P. Germonpré, M. Huizing, V. Van Tendeloo, K. Saevels, L. Rutsaert, K. Vermeulen, A. Snoeckx, B. Op de Beeck, N. Cools, G. Nijs, B. Stein, E. Lion, A. van Driessche, M. Peeters, E. Smits. Vaccination of cancer patients with dendritic cells electroporated with mRNA encoding the Wilms' Tumor protein (WT1): correlation of clinical effect and overall survival with T-cell response. Cytotherapy 2019, 21(5), p. S10.
- [Background] Z. Berneman, A. Van de Velde, S. Anguille, Y. Willemen, M. Huizing, P. Germonpré, K. Saevels, G. Nijs, N. Cools, A. Van Driessche, B. Stein, H. De Reu, W. Schroyens, A. Gadisseur, A. Verlinden, K. Vermeulen, M. Maes, M. Lammens, H. Goossens, M. Peeters, V. Van Tendeloo, E. Smits. Vaccination with Wilms' Tumor Antigen (WT1) mRNA-Electroporated Dendritic Cells as an Adjuvant Treatment in 60 Cancer Patients: Report of Clinical Effects and Increased Survival in Acute Myeloid Leukemia, Metastatic Breast Cancer, Glioblastoma and Mesothelioma. Cytotherapy 2016, 18(6), p. S13-14
- [Derived] Shallis RM, Podoltsev NA. Maintenance therapy for acute myeloid leukemia: sustaining the pursuit for sustained remission. Curr Opin Hematol. 2021 Mar 1;28(2):110-121. doi: 10.1097/MOH.0000000000000637. PMID 33394722